CLINICAL TRIAL: NCT06502717
Title: Testing the Efficacy of Viome-designed Condition-based Supplements and Viome Precision Supplements to Improve Clinical Outcomes for Mental Health Conditions
Brief Title: Viome Precision Nutritional Programs to Improve Clinical Outcomes for Mental Health Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V211.3_v2
Record Dates: First submitted 2024-06-25; First posted 2024-07-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Issue; Depression; Anxiety
Keywords: mental health; diet; supplements; vitamins; stress
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, cohort study divided into two study arms: 1) control group (placebo), 2) precision-supplement
Who Masked: Participant
Masking Description: Once enrolled, participants are randomized into one of the two arms. The coded supplements with blinded labels are shipped to the participants. The participants are not aware of which group they are randomized into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (No Intervention): Participants who have mental health issues are randomized into this study arm. They may be provided with any combination of nutritional recommendations and supplements. Placebo capsules will contain inert or inactive ingredients. Participants may need to use a mobile app in order to participate in the trial.
- Viome's Precision Nutrition Program (VPNP) (Active Comparator): Participants who have mental health issues are randomized into this arm. They may be provided with any combination of nutritional recommendations and supplements. Participants may need to use a mobile app in order to participate in the trial.
  Interventions: Combination Product: VIOME Precision Nutrition Program

INTERVENTIONS:
Combination Product: VIOME Precision Nutrition Program — Precision supplement based on the participants microbiome sample results. Participants in this arm may have any combination of supplements, diet recommendations, and/or coaching.
  Other Names: VPNP
  Arms: Viome's Precision Nutrition Program (VPNP)

SUMMARY:
US residents who have mental health issues sign the informed consent form and are screened and enrolled for this study. Participants complete a survey upon enrollment and are randomized into one of two study arms. This study is direct to participant and will NOT utilize clinical sites.

DETAILED DESCRIPTION:
Participants who meet the eligibility criteria are randomized into any of the two study arms including: the placebo arm or the VIOME Precision Nutrition Program (VPNP) arm.

Placebo and Viome's Precision Nutrition Program include supplements, may include dietary recommendations towards improving the symptoms associated with mental health. The trial will last approximately 4 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the United States
* Females and males ages 25-75 (inclusive)
* Able to speak and read English
* No unexplained weight loss, fevers, anemia, or blood in stool
* Willing and able to follow the trial instructions, as described in the recruitment letter
* Signed and dated informed consent prior to any trial-specific procedures.
* PHQ9 score of 5-24 (inclusive)

Exclusion Criteria:

* Unwilling to change their current diet
* Prior use of Viome products or services
* Antibiotic use in the previous 4 weeks
* Pregnancy (current or planned in the next 4 months)
* < 90 days postpartum
* Breast feeding
* Active infection
* Unable or unwilling to use Viome's App on an iPhone or Android smartphone
* Significant diet or lifestyle change in the previous 1 month
* IBD diagnosis -Major psychiatric/DSM-4 disease diagnosis (e.g. Schizophrenia, Bipolar disorder, Post- traumatic Stress Disorder, Obsessive Compulsive disorder)
* Use of investigational drugs, products or devices within 1 month prior to and 4 months after the start of the trial
* Cancer therapy within the previous 1 year
* Major surgery in the last 6 months or planned in the next 4 months
* Allergies to any supplement ingredients listed in the screening survey
* Currently on a specific diet: FODMAP, KETO, PALEO
* Answered yes to the question, "In the past few weeks, have you wished you were dead or had thoughts about killing yourself?"
* Gastrointestinal disease including:

  * GI surgery except:

    * Appendectomy and benign polypectomy
* Esophagitis
* Celiac disease
* GI malignancy or obstruction
* Peptic Ulcer Disease
* Duodenal or gastric ulcer disease

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reduced PHQ-9 Score | ~4 months
  Reduced PHQ-9 score for the VPNP group compared to baseline scores.
Reduced GAD-7 Score | ~4 months
  Reduced GAD-7 score for the VPNP groups compared to baseline scores.
Reduced Perceived Stress Scale Score | ~4 months
  Reduced Perceived Stress Scale score for the VPNP group compared to baseline scores.
Increased Quality of Life Score | ~4 months
  Increased quality of life score for the VPNP group compared to baseline scores.
Correlation between microbial changes and clinical outcomes | ~4 months
  Correlation between microbial changes on the VPNP with clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States